CLINICAL TRIAL: NCT00697151
Title: Patent Foramen Ovale in Cryptogenic Stroke Study
Acronym: PICSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Shunichi Homma,MD - Principal Investigator, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6372; R01NS032525 (NIH)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Ischemic Stroke; Patent Foramen Ovale
Keywords: cerebrovascular diseases; ischemic stroke; patent foramen ovale; warfarin; aspirin; transesophageal echocardiography
MeSH Terms: conditions — Ischemic Stroke; Foramen Ovale, Patent; Cerebrovascular Disorders | interventions — Warfarin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warfarin (Active Comparator): Warfarin (target International Normalized Ratio: 1.4 to 2.8) plus placebo aspirin
  Interventions: Drug: Warfarin
- Aspirin (Active Comparator): Aspirin 325 mg plus placebo warfarin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Warfarin — Warfarin once a day, titrated to obtain an INR of 1.4 to 2.8; placebo aspirin once a day
  Other Names: Coumadin
  Arms: Warfarin
Drug: Aspirin — Aspirin 325 mg once a day; placebo warfarin once a day
  Arms: Aspirin

SUMMARY:
The study sought to assess the rate of recurrent stroke and death in stroke patients with a patent foramen ovale randomized to treatment with warfarin or aspirin. This was a multicenter study conducted at 48 U.S. Institutions.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-85
* Ischemic stroke within 30 days
* Glasgow outcome scale ≥ 3
* No contraindications to warfarin/aspirin

Exclusion Criteria:

* Basal INR > 1.4
* Post-procedural stroke
* Severe carotid atherosclerosis
* Cardioembolic stroke
* Contraindications to transesophageal echocardiography

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 1993-06; Primary Completion 2000-06 (Actual); Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Recurrent ischemic stroke and death | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shunichi Homma, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia College of Physicians and Surgeons, New York, New York, United States

REFERENCES:
- [Result] Homma S, Sacco RL, Di Tullio MR, Sciacca RR, Mohr JP; PFO in Cryptogenic Stroke Study (PICSS) Investigators. Effect of medical treatment in stroke patients with patent foramen ovale: patent foramen ovale in Cryptogenic Stroke Study. Circulation. 2002 Jun 4;105(22):2625-31. doi: 10.1161/01.cir.0000017498.88393.44. PMID 12045168
- [Result] Homma S, DiTullio MR, Sacco RL, Sciacca RR, Mohr JP; PICSS Investigators. Age as a determinant of adverse events in medically treated cryptogenic stroke patients with patent foramen ovale. Stroke. 2004 Sep;35(9):2145-9. doi: 10.1161/01.STR.0000135773.24116.18. Epub 2004 Jul 1. PMID 15232117
- [Result] Homma S, Sacco RL, Di Tullio MR, Sciacca RR, Mohr JP. Atrial anatomy in non-cardioembolic stroke patients: effect of medical therapy. J Am Coll Cardiol. 2003 Sep 17;42(6):1066-72. doi: 10.1016/s0735-1097(03)00907-0. PMID 13678932
- [Derived] Di Tullio MR, Russo C, Jin Z, Sacco RL, Mohr JP, Homma S; Patent Foramen Ovale in Cryptogenic Stroke Study Investigators. Aortic arch plaques and risk of recurrent stroke and death. Circulation. 2009 May 5;119(17):2376-82. doi: 10.1161/CIRCULATIONAHA.108.811935. Epub 2009 Apr 20. PMID 19380621